CLINICAL TRIAL: NCT02054533
Title: Prospective Cohort of Ulcerative Colitis and Crohn's Disease Patients Undergoing Surgery to Identify Risk Factors for Post-Operative Infection I
Brief Title: Study to Determine Risk Factors for Post-operative Infection in Inflammatory Bowel Disease
Acronym: PUCCINI
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 12-0899
Record Dates: First submitted 2014-01-27; First posted 2014-02-04 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Crohn's disease; Ulcerative colitis; Inflammatory bowel disease; Surgery; Anti-Tumor Necrosis Factor; Infection
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBD patients: patients with IBD undergoing intra-abdominal surgery

SUMMARY:
Understanding of how best to treat inflammatory bowel disease (IBD) has evolved over the last ten years. Evidence now suggests that the most effective therapy early in the course of Crohn's disease (CD) and ulcerative colitis (UC) involves the use of immune suppressing medications such as the anti-Tumor Necrosis Factor (anti-TNF) agents infliximab, adalimumab, and certolizumab. However, many CD and UC patients still ultimately require surgery despite the use of these medications. Side effects of the anti-TNF agents include increased risk of infections due to their effect on the immune system. Little is known about how use of these medications near the time of surgery may affect patients' risks of infection or other post-operative complications. The only available studies on this topic have given conflicting results. These studies have been limited by the fact that they have been small in size and retrospective. Retrospective studies primarily involve chart review as the method of identifying potential risk factors for infections and other complications after they have already occurred. This method limits both the type and quality of information/data that can be collected. The conflicting results have led to variance in practice patterns with regards to management of anti-TNF agents, the timing of surgery, and even the types of surgery.

By enrolling patients at the time of their surgery, collecting extensive information may be possible than previously studied on potential risk factors for both infectious and non-infectious complications following surgery. Risk factors to be studied will include individual patient characteristics, disease characteristics, surgical methods, novel characteristics of CT scans and MRIs and extensive medication exposures. The primary objective is to determine if exposure to anti-TNF agents prior to surgery increases the risk of infection post-operatively. And evaluate exposure to anti-TNF agents by both patient history of use and measurement of anti-TNF drug levels at the time of surgery. Monitoring of drug levels at the time of surgery has never been utilized in this way to evaluate the risk of anti-TNF agents in IBD. However, this has been done to assess the risk of other medications in different diseases.

If anti-TNF agents are found to pose a risk for infectious or non-infectious outcomes in IBD patients undergoing surgery, change maybe needed in the way these medications are used around the time of surgery. Additionally, by collecting comprehensive information on other potential risk factors besides medication use patients at greatest risk for bad outcomes can be identified and take protective measures when possible. The aims of this study address the CCFA challenge to better define the risks of medical and surgical therapies to improve the quality of care of IBD patients undergoing surgery.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational study designed to determine if pre-operative exposure to anti-TNF agents is an independent risk factor for post-operative infectious complications within 30 days of surgery in subjects with IBD.

Patient Assessments:

Patient assessments will occur at the Screening/Baseline Visit, Discharge Day, and 30-Day Telephone Follow-up (see Figure 1). Potential pre-operative predictors of post-operative infections will be assessed at the Screening/Baseline Visit through a brief patient interview and abstraction of medical records. Data will be entered into the electronic case report forms (eCRF). A second data abstraction will occur on the Discharge Day. At this time, all data from the day of surgery will be available including finalized operative reports, anesthesia records, and pathology. The post-operative medical record will also be reviewed for potential confounding factors related to post-operative infection (i.e. presence of central lines, foley catheters, antibiotic use, etc.). Additionally, the medical record will be reviewed for the occurrence of post-operative infection and the other non-infectious outcomes being studied. Data will be entered into the eCRF. The final assessment will occur on post-operative day 30 (within 1 week). A telephone interview will be conducted. The purpose of the interview is to assess for the occurrence of post-operative infection and non-infectious outcomes. If an infection has been identified, relevant medical records will be requested to confirm infection and abstract information pertaining to the infection. Data will be entered into the eCRF.

Assessment of Anti-TNF Exposure:

Exposure to anti-TNF agents will be defined in two different ways. The primary analysis will define anti-TNF exposure as patient report of use within 12 weeks of surgery pre-operatively. Confirmation of patient report will be through medical record abstraction. This definition of anti-TNF exposure is consistent with many of the retrospective, single center studies on post-operative infections related to IBD surgery. The 12-week cutoff point has been chosen to account for the washout of infliximab before surgery based on its half-life. However, the different anti-TNF agents have varying half-lives. Date of last administration prior to surgery will be recorded so that different cutoff points to define exposure such as 4 weeks and 8 weeks may be explored.

The secondary analysis will define anti-TNF exposure by measured peri-operative levels in patients with a history of anti-TNF use in the six months preceding surgery. Anti-TNF levels and anti-drug antibodies will be checked at two time points in patients with recent anti-TNF use. An initial level will be drawn at the screening visit, which may occur peri-operatively up to post-op day 4. A second level will be drawn anytime between post-op day 4 and post-op day 7. The serum from these blood draws will be stored at -80 Celsius until the third year of the study at which time samples will be tested for drug levels and antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older;
* Diagnosis of CD, UC, or indeterminate colitis by standard criteria;
* Patient planned to have intra-abdominal surgery or has had intra-abdominal surgery in the preceding four days;
* Ability to provide written informed consent.

Exclusion Criteria:

* Current enrollment in a clinical trial for an investigational IBD therapy;
* Surgery to repair a complication from a recent surgery (≤ 90 days);
* Inability or unwillingness to provide written informed consent;
* Any other condition which may impede competence or compliance or hinder completion of the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with IBD undergoing intra-abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 974 (Actual)
Dates: Start 2014-02; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Post-Operative Infection | up to 30 days

SECONDARY OUTCOMES:
Pouch Specific Complication | up to 30 days
  1. Anastomotic Leaks
  2. Pelvic Abscesses
  3. Pouch fistula
  4. Pouch dehiscence
Hospital re-admission | up to 30 days
Re-operation secondary to surgical complication | up to 30 days
Duration of post-operative hospitalization | up to 30 days
30 day post-operative mortality | up to 30 days
Thrombotic complication | up to 30 days
Hypomotility complication | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Sands, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (24):
- United States (24):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - The University of Chicago, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Inc., Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State College of Medicine, Hershey, Pennsylvania
  - The University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburth, Pittsburgh, Pennsylvania